CLINICAL TRIAL: NCT04508244
Title: Beta Blocker Use In Traumatic Brain Injury Based On The High-Sensitive Troponin T Status: A Randomized Controlled Trial (BBTBBT)
Brief Title: Beta Blocker Use In Traumatic Brain Injury Based On The High-Sensitive Troponin T Status
Acronym: BBTBBT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRGC-05-SI-18-293
Record Dates: First submitted 2020-07-24; First posted 2020-08-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Trauma; Brain Injuries; Stress Reaction; Beta Blockers; Troponin
Keywords: propranolol; troponin; biomarkers; myocardial injury; brain injury; trauma; qatar
MeSH Terms: conditions — Wounds and Injuries; Brain Injuries; Fractures, Stress | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blinded, placebo-controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TBI with positive troponin (Active Comparator): Patients will receive IV propranolol for 6 days
  Interventions: Drug: Propranolol
- TBI with negative troponin (a) (Placebo Comparator): Patients will receive IV placebol for 6 days
  Interventions: Drug: Placebo
- TBI with negative troponin (b) (Experimental): Patients will receive IV propranolol for 6 days
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Placebo — 12 ampoules of 1 mg placebo solution (3 ampoules/day for 2 days; 2 ampoules/day for day-3 & 4 and 1 ampoule/day for day-5 & 6.
  Arms: TBI with negative troponin (a)
Drug: Propranolol — 12 ampoules of 1 mg placebo solution (3 ampoules/day for 2 days; 2 ampoules/day for day-3 & 4 and 1 ampoule/day for day-5 & 6.
  Other Names: inderal
  Arms: TBI with negative troponin (b); TBI with positive troponin

SUMMARY:
Beta blockers (BB) play an important role in protection of end organs that are susceptible for secondary injury by the Traumatic brain injury (TBI)-induced catecholamine surge. However, use of BBs in trauma patients is not yet the standard of care which necessitates clear scientific evidence and justification to be used especially in TBI patients. The BBTBBT study aims to determine whether early administration of propranolol based on the HSTnT status will improve the outcome of mild-to-severe TBI patients. Our primary hypothesis is that BBs are effective in reducing 10 and 30-day mortality in TBI patients.BBs are effective in reducing 10 and 30-day mortality in TBI patients.

Methods/Design: The BBTBBT study is a prospective, randomized, double-blinded, placebo-controlled trial, three-arm trial of BB use in mild-to-severe TBI patients based on the HsTnT status.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) accounts for up to 30% of all injury-related deaths [1]. It also poses a significant morbidity and economic burden world-wide [2,3]. While there has been significant advances in trauma care overall, there are limited medical management options for head injury. Based on retrospective observational studies, TBI is associated with an increased risk of mortality. Some of these studies reported higher rate of mortality in TBI patients who had elevated serum troponin in comparison to those who had normal troponin, even in isolated TBI.

Few studies have evaluated the clinical significance of the release of serum cardiac troponins after trauma [4-7]. Some of these studies showed that elevated troponin could reflect the degree of severity of overall body injury, but in particular the severity of thorax trauma regardless of cardiac involvement [5,6]. Furthermore, elevated troponins were reported in acute non-traumatic head injury, including acute stroke (≈27%), and subarachnoid hemorrhage (≈20%) [4, 7]. However, the precise mechanism of elevated troponin is difficult to be determined due to the multitude of prevailing clinical circumstances which may influence troponin release. Moreover, the clinical significance and prognostic value of elevated troponins levels and immune response remain poorly explored in TBI patients. Earlier studies relied mainly on TnT or TnI and did not examine the newer high-sensitive TnT (HsTnT) which has more sensitivity and shorter time to detect myocardial damage. A recent meta-analysis showed that elevated troponins are commonly seen in critically-ill patients even in the absence of coronary artery disease [7,8,9] with a prevalence of 45% studies utilized conventional troponin assays ( TnT and TnI), [10] however, this figure reaches 62% with the use of HsTnT [11, 12]. From the therapeutic point of view, BBs use was reported to have better survival in blunt TBI patients [4, 14, 15,16]. Notably, BBs play an important role in protection of end organs that are susceptible for secondary injury by the TBI-induced catecholamine surge [4]. Upon the latter observation, the use of HsTnT test early in TBI cases may allow early stratification and therapy to possibly reduce mortality. However, this assumption needs further support through large clinical trials. Prospective studies that link the release of troponins and mortality in post-TBI patients are lacking. The use of BBs in patients with acute coronary myocardial injury is evidence-based, especially in the very early hours post myocardial injury. However, use of BBs in trauma patients is not yet the standard of care. The use of BBs needs to be clearly justified in TBI patients. Retrospectively, Salim et al [13] reported that patients with severe TBI who did not receive BBs had a mortality rate of 36% vs. 24% in those who were receiving BBs (p=0.036). Furthermore, if troponin I was elevated on admission, the hospital mortality increased to 48.5% in patients without BBs therapy vs. 22.4% in those who were using BBs (p=0.026).However, the two groups (with & without BB) were comparable for mortality, if the admission troponin values were not elevated (p=0.31). In brief, the utmost benefit in survival occurred in BBs use group based on the troponin positivity on admission. However, this study did not explain the specific underlying mechanism of troponin positivity. The BBTBBT study is a prospective, randomized, double-blinded, placebo-controlled trial, three-arm trial of BB use in mild-to-severe TBI patients based on the HsTnT status. We hypothesized that early administration of BBs has beneficial effect on the 10 and 30-day mortality in patients with mild-to-severe TBI based on the admission HsTnT status.

ELIGIBILITY:
Inclusion Criteria:

* All adults (≥18 -65 years)
* both genders
* mild-to-severe blunt TBI (head AIS 1-5 and/ GCS 4-15) patients requiring hospital admission

Exclusion Criteria:

* Patients <18 and> 65 yrs old
* penetrating trauma
* non-survivable injuries (head AIS=6 & GCS=3)
* uncontrolled bleeding on arrival to ED
* pregnant women
* prisoners
* patients with heart rate (HR) ≤70, systolic blood pressure (SBP) ≤100 mmHg (or MAP <70 mmHg) not responding to initial management or required to be maintained on vasopressors on arrival .
* Patients who will undergo hypothermia therapy,
* any penetrating injury to head, thorax or abdomen,
* history of bronchial asthma
* patients posted for emergency surgery during the first 6 hrs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 10 days
  Number of participants who died from each study arm
Mortality | 30 days
  Number of participants who died from each study arm

SECONDARY OUTCOMES:
Duration of hospital stay | 3 months
  number of days in the hospital
Functional status | 3 months
  Glasgow Outcome scale (range 1-8); higher scores mean a better outcome

OTHER OUTCOMES:
Injury severity indicators | 48 hours
  correlation between blood biomarkers and head CT scan findings

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El-Menyar, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
data sharing agreement should be signed with the MRC and legal affair at HMC

REFERENCES:
- [Background] Faul M, Xu L, Wald MM, Coronado VG. Traumatic Brain Injury in the United States: Emergency Department Visits, Hospitalizations, and Deaths. Atlanta, GA: Centers for Disease Control and Prevention, National Center for Injury Prevention and Control; 2010.
- [Background] Ma VY, Chan L, Carruthers KJ. Incidence, prevalence, costs, and impact on disability of common conditions requiring rehabilitation in the United States: stroke, spinal cord injury, traumatic brain injury, multiple sclerosis, osteoarthritis, rheumatoid arthritis, limb loss, and back pain. Arch Phys Med Rehabil. 2014 May;95(5):986-995.e1. doi: 10.1016/j.apmr.2013.10.032. Epub 2014 Jan 21. PMID 24462839
- [Background] Mock C, Lormand JD, Goosen J, Joshipura M, Peden M. Guidelines for essential trauma care. Geneva, World Health Organization, 2004. Retrieved from: http://www.who.int/violence_injury_prevention/publications/services/en/guidelines_traumacare.pdf
- [Background] Al-Otaiby MA, Al-Amri HS, Al-Moghairi AM. The clinical significance of cardiac troponins in medical practice. J Saudi Heart Assoc. 2011 Jan;23(1):3-11. doi: 10.1016/j.jsha.2010.10.001. Epub 2010 Oct 20. PMID 23960628
- [Background] Mahmood I, El-Menyar A, Dabdoob W, Abdulrahman Y, Siddiqui T, Atique S, Arumugam SK, Latifi R, Al-Thani H. Troponin T in Patients with Traumatic Chest Injuries with and without Cardiac Involvement: Insights from an Observational Study. N Am J Med Sci. 2016 Jan;8(1):17-24. doi: 10.4103/1947-2714.175188. PMID 27011943
- [Background] Edouard AR, Felten ML, Hebert JL, Cosson C, Martin L, Benhamou D. Incidence and significance of cardiac troponin I release in severe trauma patients. Anesthesiology. 2004 Dec;101(6):1262-8. doi: 10.1097/00000542-200412000-00004. PMID 15564931
- [Background] Hasanin A, Kamal A, Amin S, Zakaria D, El Sayed R, Mahmoud K, Mukhtar A. Incidence and outcome of cardiac injury in patients with severe head trauma. Scand J Trauma Resusc Emerg Med. 2016 Apr 27;24:58. doi: 10.1186/s13049-016-0246-z. PMID 27121183
- [Background] Smith A, John M, Trout R, Davis E, Moningi S. Elevated cardiac troponins in sepsis: what do they signify? W V Med J. 2009 Jul-Aug;105(4):29-32. PMID 19585902
- [Background] Lim W, Cook DJ, Griffith LE, Crowther MA, Devereaux PJ. Elevated cardiac troponin levels in critically ill patients: prevalence, incidence, and outcomes. Am J Crit Care. 2006 May;15(3):280-8; quiz 289. PMID 16632770
- [Background] Poe S, Vandivier-Pletsch RH, Clay M, Wong HR, Haynes E, Rothenberg FG. Cardiac Troponin Measurement in the Critically Ill: Potential for Guiding Clinical Management. J Investig Med. 2015 Dec;63(8):905-15. doi: 10.1097/JIM.0000000000000239. PMID 26425879
- [Background] Salim A, Hadjizacharia P, Brown C, Inaba K, Teixeira PG, Chan L, Rhee P, Demetriades D. Significance of troponin elevation after severe traumatic brain injury. J Trauma. 2008 Jan;64(1):46-52. doi: 10.1097/TA.0b013e31815eb15a. PMID 18188098
- [Background] Bukur M, Mohseni S, Ley E, Salim A, Margulies D, Talving P, Demetriades D, Inaba K. Efficacy of beta-blockade after isolated blunt head injury: does race matter? J Trauma Acute Care Surg. 2012 Apr;72(4):1013-8. doi: 10.1097/TA.0b013e318241bc5b. PMID 22491619
- [Background] Schroeppel TJ, Fischer PE, Zarzaur BL, Magnotti LJ, Clement LP, Fabian TC, Croce MA. Beta-adrenergic blockade and traumatic brain injury: protective? J Trauma. 2010 Oct;69(4):776-82. doi: 10.1097/TA.0b013e3181e981b8. PMID 20938265
- [Background] Ko A, Harada MY, Barmparas G, Thomsen GM, Alban RF, Bloom MB, Chung R, Melo N, Margulies DR, Ley EJ. Early propranolol after traumatic brain injury is associated with lower mortality. J Trauma Acute Care Surg. 2016 Apr;80(4):637-42. doi: 10.1097/TA.0000000000000959. PMID 26808028
- [Background] El-Menyar A, Asim M, Latifi R, Bangdiwala SI, Al-Thani H. Predictive value of positive high-sensitivity troponin T in intubated traumatic brain injury patients. J Neurosurg. 2018 Dec 1;129(6):1541-1549. doi: 10.3171/2017.7.JNS17675. Epub 2018 Jan 5. PMID 29303440
- [Background] El-Menyar A, Goyal A, Latifi R, Al-Thani H, Frishman W. Brain-Heart Interactions in Traumatic Brain Injury. Cardiol Rev. 2017 Nov/Dec;25(6):279-288. doi: 10.1097/CRD.0000000000000167. PMID 28984668
- [Derived] El-Menyar A, Asim M, Khan N, Rizoli S, Mahmood I, Al-Ani M, Kanbar A, Alaieb A, Hakim S, Younis B, Taha I, Jogol H, Siddiqui T, Hammo AA, Abdurraheim N, Alabdallat M, Bahey AA, Ahmed K, Atique S, Chaudry IH, Prabhu KS, Uddin S, Al-Thani H. Systemic and cerebro-cardiac biomarkers following traumatic brain injury: an interim analysis of randomized controlled clinical trial of early administration of beta blockers. Sci Rep. 2024 Aug 23;14(1):19574. doi: 10.1038/s41598-024-70470-y. PMID 39179700
- [Derived] El-Menyar A, Asim M, Bahey AA, Chughtai T, Alyafai A, Abdelrahman H, Rizoli S, Peralta R, Al-Thani H. Beta blocker use in traumatic brain injury based on the high-sensitive troponin status (BBTBBT): methodology and protocol implementation of a double-blind randomized controlled clinical trial. Trials. 2021 Dec 7;22(1):890. doi: 10.1186/s13063-021-05872-8. PMID 34876207